CLINICAL TRIAL: NCT07178301
Title: Elective Neck Dosing in Low Risk Oropharyngeal Human Papillomavirus-Related Cancer Treatment (ENLIGHT): A Single Arm Prospective Phase II Assessing 30 Gy Elective Neck Dose
Brief Title: Evaluating a Decreased Dose of Radiation Therapy to the Elective Neck for the Treatment of HPV-Related Oropharyngeal Cancer, ENLIGHT Trial
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 25N01; NCI-2025-06273 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00224657; NU 25N01 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Clinical Stage I HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage II HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Magnetic Resonance Spectroscopy; Radiotherapy; Radiation

STUDY DESIGN:
Intervention Model Description: Patients will undergo standard of care treatment with definitive radiotherapy, to a dose of 70 Gy to gross tumor (per standard of care) and 30 Gy to the elective neck.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (radiation therapy) (Experimental): Patients receive standard dose radiation therapy to the tumor and reduced dose radiation therapy to the elective neck lymph nodes five days per week for a total of 35 fractions over 7 weeks. Patients also undergo CT, PET, and nasopharyngolaryngoscopy throughout the trial.
  Interventions: Procedure: Computed Tomography; Procedure: Nasopharyngeal Laryngoscopy; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Radiation: Radiation Therapy

INTERVENTIONS:
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Nasopharyngeal Laryngoscopy — Undergo nasopharyngolaryngoscopy
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This clinical trial evaluates how decreasing the dose of radiation to the elective neck (areas of lymph nodes not directly involved in the cancer) impacts treatment outcomes in patients with human papillomavirus (HPV)-related oropharyngeal cancer. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill cancer cells and shrink tumors. Radiation therapy plays an important role in the treatment of HPV-related oropharyngeal cancer, but it also causes significant toxicities. Given the significant toxicities associated with treatment, and the excellent outcomes of HPV-related oropharyngeal cancer, researchers are attempting to identify methods to de-escalate treatment for HPV-related oropharyngeal cancer in an effort to maintain excellent treatment outcomes while reducing the risk of toxicities. Reducing the dose of radiation therapy to the lymph nodes in the neck that aren't directly involved in the cancer may improve patient quality of life while still maintaining excellent rates of cure of disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine 2-year locoregional progression free survival (LRPFS).

SECONDARY OBJECTIVES:

I. To determine 2-year progression free survival (PFS). II. To determine 2-year regional failure in the low-dose elective region. III. To determine 2-year overall survival (OS). IV. To determine physician-reported toxicities at 1, 3, 12-months as measured by Common Terminology Criteria for Adverse Events (CTCAE).

V. To assess patient-reported toxicities at 1, 3, 12-months as measured by Functional Assessment of Cancer Therapy - Head & Neck Radiotherapy Index (FACT-HN-Rad).

OUTLINE:

Patients receive standard dose radiation therapy to the tumor and reduced dose radiation therapy to the elective neck lymph nodes five days per week for a total of 35 fractions over 7 weeks. Patients also undergo computed tomography (CT), positron emission tomography (PET), and nasopharyngolaryngoscopy throughout the trial.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed HPV-related OPSCC, confirmed by HPV in-situ hybridization
* Patients must not have received prior treatment (i.e., no induction chemotherapy)
* Patients must have evaluable disease (per Response Evaluation Criteria in Solid Tumors [RECIST] version [v]1.1 response criteria)
* Patients must be age >= 18 years
* Patients must have American Joint Committee on Cancer (AJCC) 8th edition stage I-II disease, as defined by a T-classification of T1-3, and N-classification of N1-2, without metastases (M0), as defined by physical examination (including nasopharyngolaryngoscopy) and positron emission tomography (PET)
* Patient must receive a staging PET scan prior to registration on study
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Patients may be planned to undergo radiation therapy (RT) alone or RT with concurrent chemotherapy, with chemotherapy managed at the discretion of the treating medical oncologist per standard of care
* RT is known to be teratogenic to a developing human fetus. For this reason, patients of child-bearing potential (POCBP) must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) from time of informed consent, for the duration of study participation (while actively receiving RT). Should a patient become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

  * NOTE: A POCBP is any patient (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy
    * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* POCBP must have a negative pregnancy test prior to CT simulation or sign the Department of Radiation Oncology's pregnancy testing declination form

  * Note: the timing of the pregnancy test/declination form will follow the policy of the Department of Radiology and Oncology, which requires completion of pregnancy testing or signed pregnancy declination prior to CT simulation
* Patients must have the ability to understand and the willingness to sign a written informed consent document prior to registration

Exclusion Criteria:

* Patients with cT4, cN3, or cM1 disease by AJCC 8th edition
* Patients who have had prior RT to the head/neck region that would result in overlap of RT fields
* Patients who have had prior major surgery to the head/neck region that could disrupt lymphatic flow
* Patients who have an uncontrolled intercurrent illness that would interfere with the receipt of RT including, but not limited to any of the following, are not eligible:

  * Uncontrolled connective tissue disorders (e.g. lupus, scleroderma) given potential for this to interfere with RT
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03-20 (Estimated); Primary Completion 2030-03-20 (Estimated); Study Completion 2031-03-20 (Estimated)

PRIMARY OUTCOMES:
2-year locoregional progression free survival | From the beginning of radiation therapy to the first incidence of local recurrence, regional recurrence in the neck, or death, assessed at 2 years post-treatment
  Response Evaluation Criteria in Solid Tumors version 1.1 will be used to assess tumor response. The 2-year progression free survival (PFS) estimate will be reported along with the confidence interval. Log-rank tests will be used to compare PFS across predefined subgroups. Cox proportional hazards models will be applied to assess the impact of covariates such as age, sex, baseline disease severity on PFS, when appropriate.

SECONDARY OUTCOMES:
2-year PFS | From the beginning of radiation therapy to the first incidence of local recurrence, regional recurrence in the neck, distant metastasis, or death, assessed at 2 years post-treatment
  Will be analyzed using the Kaplan-Meier method. Differences in survival distributions across patient subgroups will be evaluated using log-rank tests, and Cox models will be used to explore the effects of demographic and clinical variables on PFS.
2-year regional failure in the low-dose elective neck region | At 2 years post-treatment
2-year overall survival (OS) | From the beginning of radiation therapy to death from any cause, assessed at 2 years post-treatment
  Will be analyzed using the Kaplan-Meier method. Log-rank tests and Cox proportional hazards models may be used to explore differences in OS by covariates such as age, sex, and baseline disease severity when appropriate.
Incidence of physician-reported adverse events (AEs) | At 1, 3, and 12 months post-treatment
  Will be measured by Common Terminology Criteria for Adverse Events version 5.0. Will generate adverse event summaries, which will include maximum grade, attribution, and frequency, based on the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. AEs will be graded as mild, moderate, severe, or life-threatening. All reported toxicities will be summarized by toxicity type and maximum grade, and sorted by the number of patients experiencing each toxicity. For each patient, the maximum grade of a given toxicity will be determined across all timepoints. AE data will be presented using categorical analyses and descriptive summary statistics. No formal statistical hypothesis testing will be performed.
Incidence of patient-reported adverse events | At 1, 3, and 12 months post-treatment
  Will be measured by Functional Assessment of Cancer Therapy - Head & Neck Radiotherapy Index.

CONTACTS AND LOCATIONS:
Overall Officials: Laila A Gharzai, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States